CLINICAL TRIAL: NCT01622101
Title: Acute Effects of Zantrex-3 on Energy Expenditure and Appetite Sensations
Brief Title: Thermogenic Properties of Zantrex-3
Acronym: ZANTREX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, AAstrup, Professor, Dr Med, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B238
Record Dates: First submitted 2012-06-14; First posted 2012-06-18 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Obesity
Keywords: Energy expenditure; Appetite; Bioactive herbal compounds; blood pressure
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- zantrex (Experimental): The test compound was administered as tablets. The Zantrex-3® compound contained yerba maté, caffeine, guarana, damiana, green tea, kola nut, schizonepeta, piper nigrum, ginseng, maca root, and cocoa nut. The content of xantines (caffeine and caffeine-like stimulants) accounted for 365 mg per serving (2 capsules).
  Interventions: Dietary Supplement: Thermogenic properties of Zantrex-3®
- Control (Placebo Comparator): The placebo supplement contained rice flower and could not be distinguished from the Zantrex-3® compound with regard to colour, taste, smell or appearance.
  Interventions: Dietary Supplement: Thermogenic properties of Zantrex-3®

INTERVENTIONS:
Dietary Supplement: Thermogenic properties of Zantrex-3® — The present study was designed as a 2-arm randomised, placebo-controlled, double-blind crossover study. Each treatment was separated by >7 d washout period. Both treatments were administered as tablets. The Zantrex-3® compound contained yerba maté, caffeine, guarana, damiana, green tea, kola nut, schizonepeta, piper nigrum, ginseng, maca root, and cocoa nut. The content of xantines (caffeine and caffeine-like stimulants) accounted for 365 mg per serving (2 capsules) or 1095 mg (6 capsules) if given as a daily dose. The placebo supplement contained rice flower and could not be distinguished from the Zantrex-3® compound with regard to colour, taste, smell or ap-pearance.

SUMMARY:
Background: Zantrex-3® is a popular dietary supplement for weight control, which consists of a combination of yerba mate, guarana, caffeine and damiana. The combination has previously been shown to decrease gastric emptying and its weight controlling effects may be related to increased satiety and thermogenesis.

Objective: To investigate the effect of Zantrex-3® on energy expenditure, hemodynamic factors and subjective appetite sensations.

Design: Twenty-three men (BMI: 23.9±3.2 kg/m2, mean±SD) participated in a randomized, double-blind, placebo-controlled crossover study. The Zantrex-3® compound contained 365 mg xantines (caffeine and caffeine-like stimulants), yerba mate, guarana and damiana. The thermogenic effect was measured for 3 hours post-intake. Blood pressure (BP), heart rate (HR) and appetite ratings were assessed every half hour.

ELIGIBILITY:
Inclusion Criteria:

* Healthy,
* BMI: 23-30 kg/m2,
* Weight stable (within +/- 3 kg) two months prior to study inclusion,
* Non-smoking,
* Nonathletic (< 10 h hard physical activity), *The subjects followed a normal Danish habitual diet with rare use of hot spices

Exclusion Criteria:

* Change in smoking status,
* Daily or frequent use of medication,
* Suffering from metabolic diseases,
* Suffering from psychiatric diseases,
* Suffering from any other clinical condition, which would make the subject unfit to participate in the study,

  * use of dietary supplements or frequent use of medication
  * blood pressure above 160/90 mmHg

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2007-05; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Acute 3-h changes from baseline in energy expenditure and respiratory quotient (RQ) | Measured on 2 seperate test days in a crossover design. Each test day is seperated by >7 days.respiratory measurements were of 3-h duration post dose
  Subjects underwent assessments of resting metabolic rate (RMR) and respiratory quotient (RQ) by indirect calorimetry using a ventilated hood system (Oxycon Champion, Mijnhardt B.V, Bunnick, The Nederlands).
  The respiratory measurements were of 3-h duration; from 10 a.m. to 1 p.m. Two baseline measurements (25 minutes) were performed between 9 a.m - 10 a.m. At 10 a.m the participants ingested one serving of the Zantrex-3® supplement or placebo and 25-minutes respiratory measurements were repeated 6 times over the next 3 hours (post-dose).

SECONDARY OUTCOMES:
3-h acute change in blood pressure (systolic and diastolic) | Measured on 2 seperate test days in a crossover design. Each test day is seperated by >7 days. Measurements were carried out at baseline and time 30, 60, 90, 120, 150 and 180 minutes
  Heart rate and blood pressure were measured using a digital blood pressure meter with an automati-cally inflating cuff of appropriate cuff size. The results were given as means of 2 to 3 consecutive measurements
3-h acute change in heart rate | Measured on 2 seperate test days in a crossover design. Each test day is seperated by >7 days. Measurements were carried out at baseline and time 30, 60, 90, 120, 150 and 180 minutes
  Heart rate and blood pressure were measured using a digital blood pressure meter with an automati-cally inflating cuff of appropriate cuff size. The results were given as means of 2 to 3 consecutive measurements
Acute 3-h changes from baseline in subjective appetite sensations using visual analogue scales | Measured on 2 seperate test days in a crossover design. Each test day is seperated by >7 days. On each test day appetite sensations are measured prior to the test compound (time 0) and 30, 60, 90, 120, 150, 180 minutes post intake
  Assessment of subjective appetite sensations (visual analogue scales (VAS)) at time 0 (baseline - prior to the test meal) and at time 15, 30, 45, 60, 90, 120, 150, 180 minutes post intake.
  Measured subjective appetite sensations of hunger, satiety, prospective consumption, fullness, composite appetite score and sensory desires to something sweet, salty, rich in fat, or meat/fish.
Acute 3-h changes from baseline in self-reported discomfort | Measured on 2 seperate test days in a crossover design. Each test day is seperated by >7 days. On each test day the subjects were asked if they felt any physiological discomfort after ingesting the test compound
  The subjects were asked about physiological discomfort trought out the test days.

CONTACTS AND LOCATIONS:
Overall Officials: Arne Astrup, Professor, Dr Med, Principal Investigator — Department of Human Nutrition, Faculty of Science, University of Copenhagen, Denmark
Locations (1):
- Department of Human Nutrition, Faculty of Science, University of Copenhagen, Denmark, Frederiksberg, Denmark